CLINICAL TRIAL: NCT02322515
Title: The Effect of a Patellar Taping on Proprioceptive Exercises in Young Women With Patellofemoral Pain Syndrome: A Single-blinded Randomized Controlled Trial.
Brief Title: Patellar Taping on Proprioceptive Exercises in Young Women With Patellofemoral Pain Syndrome
Acronym: Tapping
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Norte do Paraná (Other)
Collaborators: Universidade Estadual de Londrina (Other)
Responsible Party: Principal Investigator, Rubens Alexandre da Silva Jr, Titular professor, Universidade Norte do Paraná
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Unopar-Rubens
Record Dates: First submitted 2014-12-15; First posted 2014-12-23 (Estimated); Last update posted 2015-12-02 (Estimated); Status verified 2015-11

CONDITIONS: Anterior Knee Pain Syndrome
Keywords: Knee; Proprioception; Electromyography; Taping
MeSH Terms: conditions — Patellofemoral Pain Syndrome

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intervention Taping (Experimental): The experimental group will use a rigid patellar taping (G1, n = 22) for the correction of lateralization of the patella and stabilization of the knee. The lateral stabilization will be made with self-adhesive taping positioned in the lateral border of the patella and tensioned in relation to the medial portion of the femur condyle, which allows an edge of the medial board patella and a stretching of lateral structures of the knee. All procedure will follow the recommendation from McConnell studies with regard to the patellar femoral syndrome.
  Interventions: Other: Intervention taping
- Placebo Taping (Placebo Comparator): The placebo group will use a rigid patellar taping (G2, n = 22), but without no correction of lateralization of the patella and/or stabilization of the knee. The taping will be placed incorrectly such as in the vertical position of knee and without any tension or traction around structures and patella.
  Interventions: Other: Placebo Taping

INTERVENTIONS:
Other: Intervention taping — A rigid patellar taping will be used for the correction in lateralization of the patella and more stabilization of the knee.
  Other Names: Patellar taping
  Arms: Intervention Taping
Other: Placebo Taping — A rigid patellar taping will be used in the vertical position and without no correction in lateralization of the patella and/or stabilization of the knee.
  Other Names: Sham taping
  Arms: Placebo Taping

SUMMARY:
The relevance of this study is to determine the effects of a patellar taping on muscle activation of the vastus medialis oblique (VMO), vastus lateralis (VL) and gluteus medius (GM) during different proprioceptive exercises frequently utilized in rehabilitation program.

DETAILED DESCRIPTION:
The purpose of this study is to assess the role of the patellar taping on muscle activation during seven proprioceptive exercises in women with the patellofemoral pain syndrome.

Forty voluntary young women (from 18 to 35 years) with three or more clinical symptoms of patellofemoral pain syndrome will be recruited. The participants will answer a clinical questionnaire in regard to knee pain and a specific patellofemoral questionnaire titled: the Anterior Knee Pain Scale (AKPS). All participants will sign an informed consent form approved by the North of Parana University Ethics Committee for Research on Human Subjects. The sample will be randomized in two groups: (G1) the experimental group that will use a rigid patellar taping (n = 20) for the correction in lateralization of the patella and stabilization of the knee. The lateral stabilization will be made with self-adhesive taping positioned in the lateral border of the patella and tensioned in relation to the medial portion of the femur condyle, which allows an edge of the medial board patella and a stretching of lateral structures of the knee. All procedure will follow the recommendation from McConnell studies with regard to the patellar femoral syndrome; and (G2) the placebo group that will use a rigid patellar taping (n = 20), but without no correction of lateralization of the patella and/or stabilization of the knee. The taping will be placed incorrectly such as in the vertical position of knee and without any tension or traction around structures and patella. A computer will be used to generate the randomization sequence of the participants. The allocation will be printed in cards by sequentially numbered in opaque envelopes.

Before performing the exercises, a maximum voluntary isometric contraction will be performed for the knee extensor muscles (e.g. specifically the VMO and VL) and hip abductor muscles (e.g. GM) in order to normalize the signal EMG for determining of the level muscular activity during each exercise, with the correct taping and/or placebo. All participants, after randomization, will perform seven proprioceptive exercises on one leg-stance position in different surfaces: 1) static position in force platform, 2) dynamic in flexion-extension knee on a force platform, 3) anteroposterior sway on rectangular rocker board, 4) mediolateral sway on rectangular rocker board, 5) unipodal standing on a swing apparatus, 6) unipodal standing on a mini-trampoline, and 7) unipodal standing on bosu balance ball. Each exercise has a time of 15 seconds performance, while sway centre of pressure parameters will be computed (exercise #1 and #2), and EMG surface will recording (VMO, VL, GM) for all seven. First, one baseline measure (without taping) will be performed and immediately after with the use of taping (intervention or placebo).

An ANOVA two-way will be performed to compare the two groups (G1 and G2) and two times (before and immediately after with taping) and the effects of interaction (Groups x Times). The size effect also will be computed to determine the rate of the changes observed.

ELIGIBILITY:
Inclusion Criteria:

* anterior or retropatellar knee pain on at least two of the following activities: prolonged sitting, stairs, squatting, running, kneeling, and hopping/jumping,
* pain on patellar palpation,
* pain while stepping down from a 25-cm step or during a double leg squat,
* symptoms for at least 1 month, average pain level of 3 cm or more on a 10-cm VAS.

Exclusion Criteria:

* signs or symptoms of other pathology including coexisting pathology, a recent history (within 3 months) of knee surgery,
* history of patellar dislocation/subluxation, or clinical evidence of meniscal lesion, ligamentous instability, traction, apophysitis around the patellofemoral complex, patellar tendon pathology, chondral damage, osteoarthritis, or referred pain from the spine, features that could affect the implementation of the trial,
* previous experience with patellar taping, an inability to attend a physical therapy clinic for a 6-wk treatment program,
* allergic reaction to adhesive tape,
* pregnancy, and an inability to understand the experimental protocol.

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2015-01; Primary Completion 2015-07 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Muscular activation level (EMG measures) | Baseline and immediately after with the taping
  Surface EMG signals will be record in the the vastus medialis oblique (VMO), vastus lateralis (VL) and gluteus medius (GM) muscles, before and immedialty after with taping, during seven proprioceptive exercises.

SECONDARY OUTCOMES:
Postural control measures (force platform) | Baseline and immediately after with the taping
  Stabilographic analysis of COP data from the force platform will used for the calculation of the main balance parameters of postural instability (ellipse area of COP and velocity sway of COP in both antero-posterior and medio-lateral directions of movement.

CONTACTS AND LOCATIONS:
Overall Officials: Rubens A DA SILVA, PhD, Principal Investigator — Universidade Norte do Paraná

REFERENCES:
- [Background] Cowan SM, Bennell KL, Crossley KM, Hodges PW, McConnell J. Physical therapy alters recruitment of the vasti in patellofemoral pain syndrome. Med Sci Sports Exerc. 2002 Dec;34(12):1879-85. doi: 10.1097/00005768-200212000-00004. PMID 12471291
- [Background] McCONNELL J. The management of chondromalacia patellae: a long term solution. Aust J Physiother. 1986;32(4):215-23. doi: 10.1016/S0004-9514(14)60654-1. PMID 25025219
- [Background] Lee SE, Cho SH. The effect of McConnell taping on vastus medialis and lateralis activity during squatting in adults with patellofemoral pain syndrome. J Exerc Rehabil. 2013 Apr;9(2):326-30. doi: 10.12965/jer.130018. Epub 2013 Apr 25. PMID 24278879
- [Derived] Araujo CG, de Souza Guerino Macedo C, Ferreira D, Shigaki L, da Silva RA. Mcconnell's patellar taping does not alter knee and hip muscle activation differences during proprioceptive exercises: A randomized placebo-controlled trial in women with patellofemoral pain syndrome. J Electromyogr Kinesiol. 2016 Dec;31:72-80. doi: 10.1016/j.jelekin.2016.09.006. Epub 2016 Sep 21. PMID 27693990